CLINICAL TRIAL: NCT01694914
Title: Comparative Study of Two Corneal Graft Storage Media: New Animal Compound Free Medium Versus Reference Medium
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0908018; 2010-A00234-35 (Other: AFSSAPS)
Record Dates: First submitted 2012-09-25; First posted 2012-09-27 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Corneal Transplantation
Keywords: Corneal Transplantation; corneal organ culture medium; free animal compound medium
MeSH Terms: interventions — Corneal Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Animal Compound Free Medium (Experimental): Patients in this arm receive a corneal graft stored in organ culture in a animal compound free medium
  Interventions: Procedure: corneal graft
- organ culture medium containing 2% of fœtal calf serum (Active Comparator): Patients in this arm receive a corneal graft stored in organ culture in a commercial organ culture medium containing 2% of fœtal calf serum
  Interventions: Procedure: corneal graft

INTERVENTIONS:
Procedure: corneal graft

SUMMARY:
At present, all commercially available corneal organ culture media contain foetal calf serum (FCS) and sometimes other compounds extracted from animals. These compounds are necessary for corneal cell survival but are problematic because they theoretically have risk of anthropozoonosis transmission, especially for new variant of CJD and the variability between FCS batches influence graft quality. Our laboratory research allowed in vitro and ex vivo validation of a new medium free compound animal. We proved its superiority over conventional medium containing 2% FCS for endothelial cell survival during the storage time. The goal of this clinical trial is now to assess its superiority in patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* over 18 years of age
* Clinically proven corneal disease
* Registered on the French National waiting list (GLAC)
* Patient informed consent
* Patient who needs a 8.25mm of diameter perforating keratoplasty, either isolated or combined with lens surgery
* Low immune rejection risk (< 2 quadrants of neovascularization, no previous history of herpetic keratitis nor graft rejection)
* No previous history of glaucoma or elevated intra ocular pressure (>22 mm

Exclusion Criteria:

* Patient is unlikely to comply with the requirements of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2012-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
the primary outcome is the endothelial cell density (ECD) of the corneal grafts. | one year after graft

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Thuret, MD-PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (4):
- France (4):
  - CHU Besançon, Besançon
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Grenoble, Grenoble
  - CHU Saint-Etienne, Saint-Etienne